CLINICAL TRIAL: NCT06079671
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multi-centre, Global Study of Volrustomig in Women With High Risk Locally Advanced Cervical Cancer Who Have Not Progressed Following Platinum-based, Concurrent Chemoradiation Therapy (eVOLVE-Cervical)
Brief Title: Study of Volrustomig in Women With High Risk Locally Advanced Cervical Cancer (eVOLVE-Cervical)
Acronym: eVOLVECervical
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Gynecologic Oncology Group Foundation (Unknown); European Network for Gynaecological Oncological Trial Groups (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D7984C00002; GOG-3092 (Other: Gynecologic Oncology Group Foundation); ENGOT-cx19/GEICO (Other: European Network for Gynaecological Oncological Trial groups); 165663 (Registry Identifier: FDA-IND); 2023-504374-38-00 (Other: EU CT)
Record Dates: First submitted 2023-09-04; First posted 2023-10-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Locally Advanced Cervical Cancer
Keywords: Locally Advanced Cervical Cancer;; Adolescent and Young Adult;; Volrustomig
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Volrustomig (Experimental): Volrustomig
  Interventions: Biological: Volrustomig
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Volrustomig — IV Infusion
  Arms: Volrustomig
Other: Placebo — IV Infusion
  Other Names: Saline
  Arms: Placebo

SUMMARY:
This is a phase III, randomized, double-blind, placebo-controlled, multi-center, global study to explore the efficacy and safety of volrustomig in women with high-risk LACC (FIGO 2018 stage IIIA to IVA cervical cancer) who have not progressed following platinum-based CCRT.

DETAILED DESCRIPTION:
Women with locally advanced cervical cancer will be randomized in a 1:1 ratio to receive treatment with Volrustomig or Placebo.

ELIGIBILITY:
Inclusion Criteria:

For inclusion in the study, patients should fulfill the following criteria:

1. Female.
2. Aged at least 15 years at the time of screening. Note: Participants < 18 years of age: physical changes should be aligned with Tanner Stage III.
3. Body weight > 35 kg.
4. Histologically documented FIGO 2018 Stage IIIA to IVA cervical adenocarcinoma, cervical squamous carcinoma, or cervical adenosquamous carcinoma, with no evidence of metastatic disease.
5. Initial staging procedures performed no more than 56 days prior to the first dose of CCRT.
6. Provision of FFPE tumor sample to assess the PD-L1 expression.
7. Must not have progressed following CCRT, participants with persistent disease after definitive CCRT must not be amenable to other available therapies with curative intent.
8. WHO/ECOG performance status of 0 or 1; duration of life expectancy of ≥ 12 weeks.
9. Adequate organ and bone marrow function.
10. Capable of providing signed informed consent.

Exclusion Criteria:

Patients should not enter the study if any of the following exclusion criteria are fulfilled:

1. Diagnosis of small cell (neuroendocrine) or mucinous adenocarcinoma of cervical cancer.
2. Evidence of metastatic disease.
3. Intent to administer a fertility-sparing treatment regimen.
4. History of organ transplant or allogenic stem cell transplant.
5. History of active primary immunodeficiency or active or prior documented autoimmune or inflammatory disorders.
6. Uncontrolled intercurrent illness.
7. History of another primary malignancy except for a) Malignancy treated with curative intent with no known active disease ≥2 years before the first dose of study intervention; b) Adequately treated nonmelanoma skin cancer or lentigo maligna, or carcinoma in situ without evidence of disease.
8. Unresolved toxicities from previous CCRT except for irreversible toxicity that is not reasonably expected to be exacerbated.
9. Prior history or presence of vesicovaginal, colovaginal, or rectovaginal fistula.
10. History of anaphylaxis to any biologic therapy or vaccine.
11. Current or prior use of immunosuppressive medication within 14 days before the first dose of the study intervention is excluded. The following are exceptions to this criterion: a) Intranasal, inhaled, topical steroids, or local steroid injections (eg, intraarticular injection); b) Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication or chemotherapy premedication) or a single dose for palliative purpose (eg, pain control); c) Physiologic doses of oral corticosteroids, ie, not exceeding 10 mg/day of prednisone (or equivalent) in the preceding 14 days.
12. Patients who have undergone a previous hysterectomy, including a supracervical hysterectomy, or will have a hysterectomy as part of their initial cervical cancer therapy.
13. Any prior (besides prior CCRT) or concurrent treatment for cervical cancer.
14. Major surgical procedures within 4 weeks prior to the first dose of the study intervention or still recovering from prior surgery.
15. Exposure to immune mediated therapy prior to the study for any indication.
16. Receipt of live attenuated vaccine within 30 days prior to the first dose of the study intervention.
17. Participants with a known allergy or hypersensitivity to the study intervention, or any excipients of the study intervention.

Min Age: 15 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 800 (Estimated)
Dates: Start 2023-09-22 (Actual); Primary Completion 2027-11-26 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) based on the investigator assessment in all randomized participants (FAS) | Up to approximately 7 years
  PFS is defined as the time from date of randomization until RECIST 1.1- defined radiological progression or histopathologically confirmed progression as assessed by the Investigator or death due to any cause, whichever occurs earlier.

SECONDARY OUTCOMES:
Overall Survival (OS) in all randomized participants | Up to approximately 7 years
  OS defined as time from randomization until the date of death due to any cause.
Objective Response Rate (ORR) in all randomized participants | Up to approximately 7 years
  ORR is defined as the proportion of participants who have a CR or PR, as determined by Investigator per RECIST 1.1
Duration of Response (DoR) in all randomized participants | Up to approximately 7 years
  DoR in participants with a CR or PR: Time from date of first detection of CR or PR until the date of RECIST 1.1-defined radiological progression or histopathologically confirmed progression.
Time to First Subsequent Therapy or death (TFST) in all randomized participants | Up to approximately 7 years
  TFST: The time from randomization until the start date of the first subsequent anti-cancer therapy after discontinuation of randomized treatment, or death due to any cause.
Time to second progression or death (PFS2) in all randomized participants | Up to approximately 7 years
  PFS2: The time from randomization to the earliest of the progression event (following the initial Investigator-assessed progression), after first subsequent therapy, or death. The date of second progression will be recorded by the Investigator in the eCRF and defined according to local standard clinical practice.
PFS by BICR in all randomized participants | Up to approximately 7 years
  Endpoints based on the PFS by BICR assessment according to RECIST 1.1.
The incidence of local progression, and distant disease progression as the first documented progression event in all randomized participants | Up to approximately 7 years
  Incidence of Local Progression, and Distant Disease Progression: Number and percentage of participants who develop local progression, distant disease recurrence.
PK of volrustomig | Up to approximately 7 years
  Concentration of volrustomig in serum and PK parameters as data allow.
The immunogenicity of volrustomig | Up to approximately 7 years
  Incidence of ADAs against volrustomig in serum.
Incidence of adverse events of volrustomig compared to placebo | Up to approximately 7 years
  An AE is defined as the development of any untoward medical occurrence (other than progression of the malignancy under evaluation) in a patient or clinical study participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment.
Participant-reported disease-related symptoms | Up to approximately 7 years
  Change from baseline as measured by the European Organization for Research and Treatment of Cancer IL318 (EORTC IL318, Symptom Experience subscale of the EORTC Quality of Life Questionnaire Symptom Specific Scale for Cervical Cancer (EORTC QLQ-CX24)). The score of scale for EORTC IL318 is from 1-4.
Participant-reported physical functioning | Up to approximately 7 years
  Change from baseline of physical functioning as measured by the Patient Reported Outcomes Measurement Information System - Short Form - Physical Functioning 8c (PROMIS SF-PF 8c). The score of scale for PROMIS SF-PF 8c is from 1-5.
Participant-reported global health status/Quality of Life | Up to approximately 7 years
  Change from baseline of Global Health Status/ Quality of Life (GHS/QoL) as measured by the European Organization for Research and Treatment of Cancer IL172 (EORTC IL172). The score of scale for EORTC IL172 is from 1-7.

CONTACTS AND LOCATIONS:
Locations (159):
- United States (27):
  - Research Site, Birmingham, Alabama
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Little Rock, Arkansas
  - Research Site, La Jolla, California
  - Research Site, West Hollywood, California
  - Research Site, Atlanta, Georgia
  - Research Site, Augusta, Georgia
  - Research Site, Savannah, Georgia
  - Research Site, Melrose Park, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, New Orleans, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, New York, New York
  - Research Site, Syracuse, New York
  - Research Site, Cleveland, Ohio
  - Research Site, Columbus, Ohio
  - Research Site, Eugene, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Providence, Rhode Island
  - Research Site, Dallas, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Fairfax, Virginia
  - Research Site, Richmond, Virginia
- Brazil (12):
  - Research Site, Barretos
  - Research Site, Belo Horizonte
  - Research Site, Curitiba
  - Research Site, Fortaleza
  - Research Site, Natal
  - Research Site, Porto Alegre
  - Research Site, Porto Velho
  - Research Site, Recife
  - Research Site, Rio de Janeiro
  - Research Site, Salvador
  - Research Site, São Paulo
  - Research Site, Teresina
- Canada (5):
  - Research Site, Hamilton, Ontario
  - Research Site, London, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Ste-Foy, Quebec
- China (26):
  - Research Site, Beijing
  - Research Site, Changde
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Chongqing
  - Research Site, Fuzhou
  - Research Site, Ganzhou
  - Research Site, Guangzhou
  - Research Site, Hangzhou
  - Research Site, Harbin
  - Research Site, Kunming
  - Research Site, Lanzhou
  - Research Site, Linyi
  - Research Site, Luzhou
  - Research Site, Nanchang
  - Research Site, Shandong
  - Research Site, Shanghai
  - Research Site, Shenyang
  - Research Site, Shenzhen
  - Research Site, Tianjin
  - Research Site, Wuhan
  - Research Site, Xi'an
  - Research Site, Yibin
  - Research Site, Yinchuan
  - Research Site, Zhengzhou
  - Research Site, Zhuzhou
- Denmark (3):
  - Research Site, Aarhus N
  - Research Site, København Ø
  - Research Site, Odense
- Germany (4):
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Hamburg
  - Research Site, Leipzig
- India (9):
  - Research Site, Calicut
  - Research Site, Jaipur
  - Research Site, Lucknow
  - Research Site, Madurai
  - Research Site, Mohali
  - Research Site, Nagpur
  - Research Site, Nashik
  - Research Site, New Delhi
  - Research Site, Vadodara
- Italy (11):
  - Research Site, Bari
  - Research Site, Bologna
  - Research Site, Catania
  - Research Site, Florence
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Monza
  - Research Site, Napoli
  - Research Site, Roma
  - Research Site, Rome
  - Research Site, Turin
- Japan (16):
  - Research Site, Fukuoka
  - Research Site, Ginowan-shi
  - Research Site, Hidaka-shi
  - Research Site, Kagoshima
  - Research Site, Kōtoku
  - Research Site, Kurume-shi
  - Research Site, Maebashi
  - Research Site, Matsuyama
  - Research Site, Morioka
  - Research Site, Nagoya
  - Research Site, Osaka
  - Research Site, Sapporo
  - Research Site, Shinjuku-ku
  - Research Site, Suita-shi
  - Research Site, Sunto-gun
  - Research Site, Toon-Shi
- Mexico (7):
  - Research Site, Coyoacán
  - Research Site, Culiacán
  - Research Site, Guadalajara
  - Research Site, Guadalajra
  - Research Site, Mexico City
  - Research Site, México
  - Research Site, Monterrey
- Norway (2):
  - Research Site, Oslo
  - Research Site, Trondheim
- Peru (2):
  - Research Site, Concepción
  - Research Site, Lima
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Gliwice
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Poznan
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, San Juan, Puerto Rico
- South Korea (4):
  - Research Site, Daegu
  - Research Site, Goyang-si
  - Research Site, Gyeonggi-do
  - Research Site, Seoul
- Spain (8):
  - Research Site, A Coruña
  - Research Site, Barcelona
  - Research Site, Córdoba
  - Research Site, Girona
  - Research Site, Hospitalet deLlobregat
  - Research Site, Madrid
  - Research Site, Palma de Mallorca
  - Research Site, Valencia
- Taiwan (7):
  - Research Site, Changhua
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
  - Research Site, Taoyuan District
- Thailand (3):
  - Research Site, Bangkok
  - Research Site, Muang
  - Research Site, Udon Thani
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Karşıyaka

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/